CLINICAL TRIAL: NCT06600191
Title: Capstan Medical TMVR Study: First-in-Human Evaluation of the Capstan TMVR System
Brief Title: Capstan Medical TMVR Study: FIH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capstan Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CL_03945
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Mitral Regurgitation
Keywords: TMVR; mitral regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Implant (Experimental): Participants who pass all screening criteria will undergo a percutaneous procedure for the implantation of a permanent mitral valve replacement device.
  Participants will be followed for 5 years to evaluate safety and feasibility of Capstan Medical TMVR System for mitral valve replacement in humans with predominantly regurgitant mitral valves who are symptomatic and who are not good surgical candidates.
  Interventions: Device: Capstan System transcatheter mitral valve replacement

INTERVENTIONS:
Device: Capstan System transcatheter mitral valve replacement — This is a first human use trial exploring a novel transcatheter mitral valve replacement implant and electro-mechanical delivery system. The device offers a minimally invasive repair for patients who have at symptomatic regurgitation who are otherwise ineligable for surgical intervention, or who have no other prospects for treatment and in whom medical therapy has already been optimised.

SUMMARY:
This study is a prospective, multi-center, non-randomized first in human study to evaluate the safety and feasibility of the Capstan Medical TMVR System for intervention in adults with moderate-severe or greater mitral regurgitation who are not surgical candidates.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of consent.
* Moderate-severe (3+) or severe (4+) mitral regurgitation
* NYHA II or greater symptoms despite optimal medical treatment.
* The local multi-disciplinary heart team agrees that TMVR is the preferred treatment over surgical intervention or other available treatment options (such as TEER).
* Ability and willingness to provide written informed consent prior to any study related procedure(s).

Exclusion Criteria:

* LVEF less than 20%
* Anatomic features (e.g., annular dimensions, neo-LVOT area, transfemoral and transseptal access, excessive MAC) unsuitable for the Capstan System
* Severe aortic valve stenosis or regurgitation
* Severe mitral stenosis
* Severe right ventricular dysfunction or severe tricuspid valve disease
* Evidence of intracardiac thrombus, vegetation, or mass
* Prior mitral valve intervention that would interfere with the appropriate placement of the Capstan Valve
* Any percutaneous coronary, carotid, or other endovascular intervention within 30 days prior to procedure
* Myocardial infarction within 30 days prior to procedure
* Cardiac resynchronization therapy (CRT) device implanted within 30 days of procedure
* Active endocarditis, other ongoing infection requiring antibiotic therapy
* Stroke or transient ischemic attack (TIA) within 30 days of procedure
* Active peptic ulcer or active gastrointestinal bleeding
* Severe pulmonary arterial hypertension with fixed PASP greater than 85mmHg
* End-stage renal failure on dialysis
* Life expectancy less than 1 year
* Subject is on the waiting list for a heart transplant or has had a prior heart transplant
* Pregnant (Participants of childbearing age are required to have a negative pregnancy test).
* Known allergy to antiplatelet therapy, heparin, or to device materials
* Inability to tolerate anticoagulation or antiplatelet therapies
* Absence of appropriate venous access
* Unable to have transesophageal echocardiography
* Unwillingness to complete the required follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of procedural success | Procedure through 30 days
  Number of participants with successful valve deployment and freedom from death or re-hospitalization for heart failure at 30 days.

SECONDARY OUTCOMES:
Technical Success | 30-Days
  Technical success is defined as successful Capstan Valve deployment with none/trace or mild mitral regurgitation at 30 days post- procedure.
Freedom from MAE | 30-days, 90-days, 6-months, 1-year, then annually to 5-years
  Successful Capstan Valve Deployment with freedom from device- or procedure-related Major Adverse Events (MAE).
  MAE is a composite of the following device or procedure related outcomes:
  * All-cause mortality
  * Emergency cardiac or vascular surgery, or re-intervention
  * Myocardial Infarction
  * Stroke
  * Life-threatening bleeding

CONTACTS AND LOCATIONS:
Locations (3):
- Monash Health, Victorian Heart Hospital, Melbourne, Australia
- Pontificia Universidad Católica de Chile, Santiago, Chile
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Undecided